CLINICAL TRIAL: NCT00094029
Title: A Treatment Protocol For Patients With Gastrointestinal Stromal Tumor Who Are Ineligible For Participation In Other SU011248 Protocols And Are Refractory To Or Intolerant Of Imatinib Mesylate
Brief Title: A Treatment Protocol for Patients With Gastrointestinal Stromal Tumor (GIST) Who May Derive Benefit From Treatment With SU011248
Status: Approved for marketing | Type: Expanded Access
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A6181036
Record Dates: First submitted 2004-10-08; First posted 2004-10-11 (Estimated); Last update posted 2012-03-09 (Estimated); Status verified 2012-03

CONDITIONS: Gastrointestinal Neoplasm
MeSH Terms: conditions — Gastrointestinal Neoplasms | interventions — Sunitinib

INTERVENTIONS:
Drug: Sutent — Sutent, 25, 37.5, or 50 mg daily

SUMMARY:
The purpose of this study is to permit access to SU011248 for treatment use by patients with GIST given the following conditions: a) patients undergo screening, but are not eligible for participation in ongoing clinical studies such as A6181004; AND b) patients have GIST which standard treatments have not been able to control with acceptable toxicity AND c) patients have the potential to derive clinical benefit from treatment with SU011248.

DETAILED DESCRIPTION:
Given that an Expanded Access study does not meet the definition of a controlled clinical investigation, and as such, is not considered an applicable drug clinical trial per NIH, Basic Results for such studies are not required to be reported. Protocol A6181036 has been identified as an Expanded Access trial, and has been registered to ClinicalTrials.gov, however Basic Results will not be posted.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven Gastrointestinal Stomal Tumor (GIST) that is not amenable to standard therapy
* Undergone screening and found to be ineligible for participation in ongoing SU011248 clinical studies
* Patient judged to have potential to derive clinical benefit from SU011248 treatment by the treating physician
* Failed prior treatment with imatinib mesylate, defined as either progression of disease or significant toxicity during treatment with imatinib mesylate that precluded further treatment
* Male or Female, 18 years or older
* Resolution of all acute toxicities of prior therapies
* Adequate organ function

Exclusion Criteria:

* Symptomatic congestive heart failure, myocardial infarction, or coronary artery bypass graft in the last 6 months, or ongoing severe or unstable angina or any unstable arrhythmia requiring medication
* Symptomatic central nervous system metastases
* Serious acute or chronic illness
* Current treatment on another clinical trial
* Pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-09; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (105):
- United States (27):
  - Pfizer Investigational Site, Duarte, California
  - Pfizer Investigational Site, Pasadena, California
  - Pfizer Investigational Site, San Francisco, California
  - Pfizer Investigational Site, Santa Monica, California
  - Pfizer Investigational Site, Washington D.C., District of Columbia
  - Pfizer Investigational Site, Gainesville, Florida
  - Pfizer Investigational Site, Gainsville, Florida
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, Niles, Illinois
  - Pfizer Investigational Site, Park Ridge, Illinois
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, New Bedford, Massachusetts
  - Pfizer Investigational Site, Detroit, Michigan
  - Pfizer Investigational Site, Farmington Hills, Michigan
  - Pfizer Investigational Site, Minneapolis, Minnesota
  - Pfizer Investigational Site, Rochester, Minnesota
  - Pfizer Investigational Site, Creve Coeur, Missouri
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Buffalo, New York
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, The Bronx, New York
  - Pfizer Investigational Site, Durham, North Carolina
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Seattle, Washington
  - Pfizer Investigational Site, Madison, Wisconsin
- Pfizer Investigational Site, Burnos Aires, Argentina
- Australia (8):
  - Pfizer Investigational Site, Camperdown, New South Wales
  - Pfizer Investigational Site, Randwick, New South Wales
  - Pfizer Investigational Site, Auchenflower, Queensland
  - Pfizer Investigational Site, Bedford Park, South Australia
  - Pfizer Investigational Site, East Melbourne, Victoria
  - Pfizer Investigational Site, Nedlands, Western Australia
  - Pfizer Investigational Site, Ashford SA
  - Pfizer Investigational Site, Auchenflower QLD
- Austria (2):
  - Pfizer Investigational Site, Graz
  - Pfizer Investigational Site, Vienna
- Belgium (2):
  - Pfizer Investigational Site, Brussels
  - Pfizer Investigational Site, Leuven
- Canada (6):
  - Pfizer Investigational Site, Calgary, Alberta
  - Pfizer Investigational Site, Vancouver, British Columbia
  - Pfizer Investigational Site, Winnipeg, Manitoba
  - Pfizer Investigational Site, St. John's, Newfoundland and Labrador
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Montreal, Quebec
- Pfizer Investigational Site, Santiago, RM, Chile
- Pfizer Investigational Site, Bogota, Cundinamarca, Colombia
- Czechia (2):
  - Pfizer Investigational Site, Brno
  - Pfizer Investigational Site, Prague
- Denmark (2):
  - Pfizer Investigational Site, Aarhus C
  - Pfizer Investigational Site, Herlev
- Pfizer Investigational Site, Helsinki, Finland
- France (3):
  - Pfizer Investigational Site, Bordeaux
  - Pfizer Investigational Site, Lyon
  - Pfizer Investigational Site, Marseille
- Germany (4):
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Cologne
  - Pfizer Investigational Site, Düsseldorf
  - Pfizer Investigational Site, München
- Pfizer Investigational Site, Thessaloniki, Greece
- Hong Kong (2):
  - Pfizer Investigational Site, Happy Valley, Hong Kong
  - Pfizer Investigational Site, Hong Kong
- Pfizer Investigational Site, Budapest, Hungary
- India (3):
  - Pfizer Investigational Site, Mumbai, Maharashtra
  - Pfizer Investigational Site, New Delhi, National Capital Territory of Delhi
  - Pfizer Investigational Site, Vellore, Tamil Nadu
- Israel (2):
  - Pfizer Investigational Site, Tel Aviv
  - Pfizer Investigational Site, Tel Litwinsky
- Italy (7):
  - Pfizer Investigational Site, Candiolo (TO), Italy
  - Pfizer Investigational Site, Aviano (PN)
  - Pfizer Investigational Site, Aviano, PN
  - Pfizer Investigational Site, Bologna
  - Pfizer Investigational Site, Genova
  - Pfizer Investigational Site, Milan
  - Pfizer Investigational Site, Torino
- Mexico (2):
  - Pfizer Investigational Site, Guadalajara, Jalisco
  - Pfizer Investigational Site, Mexico City, Mexico City
- Netherlands (2):
  - Pfizer Investigational Site, Groningen, Provincie Groningen
  - Pfizer Investigational Site, Leiden
- Pfizer Investigational Site, Oslo, Norway
- Pfizer Investigational Site, Warsaw, Poland
- Pfizer Investigational Site, Singapore, Singapore
- Pfizer Investigational Site, Bratislava, Bratislava Region, Slovakia
- Pfizer Investigational Site, Seoul, South Korea
- Spain (6):
  - Pfizer Investigational Site, Barcelona, Barcelona
  - Pfizer Investigational Site, L'Hospitalet de Llobregat, Barcelona
  - Pfizer Investigational Site, Madrid, Madrid
  - Pfizer Investigational Site, Oviedo, Principality of Asturias
  - Pfizer Investigational Site, Seville, Sevilla
  - Pfizer Investigational Site, Valencia, Valencia
- Pfizer Investigational Site, Gothenburg, Sweden
- Pfizer Investigational Site, Lausanne, Switzerland
- Taiwan (2):
  - Pfizer Investigational Site, Kaohsiung Hsien
  - Pfizer Investigational Site, Taipei
- Thailand (2):
  - Pfizer Investigational Site, Ratchatawi, Bangkok
  - Pfizer Investigational Site, Bangkok
- Turkey (Türkiye) (3):
  - Pfizer Investigational Site, Ankara
  - Pfizer Investigational Site, Inciralti / Izmir
  - Pfizer Investigational Site, Istanbul
- United Kingdom (4):
  - Pfizer Investigational Site, Leeds, England
  - Pfizer Investigational Site, London
  - Pfizer Investigational Site, Manchester
  - Pfizer Investigational Site, Newcastle upon Tyne
- Pfizer Investigational Site, Caracas, Distrito Federal, Venezuela

REFERENCES:
- [Derived] Reichardt P, Kang YK, Rutkowski P, Schuette J, Rosen LS, Seddon B, Yalcin S, Gelderblom H, Williams CC Jr, Fumagalli E, Biasco G, Hurwitz HI, Kaiser PE, Fly K, Matczak E, Chen L, Lechuga MJ, Demetri GD. Clinical outcomes of patients with advanced gastrointestinal stromal tumors: safety and efficacy in a worldwide treatment-use trial of sunitinib. Cancer. 2015 May 1;121(9):1405-13. doi: 10.1002/cncr.29220. Epub 2015 Jan 13. PMID 25641662
- [Derived] Dudeck O, Zeile M, Reichardt P, Pink D. Comparison of RECIST and Choi criteria for computed tomographic response evaluation in patients with advanced gastrointestinal stromal tumor treated with sunitinib. Ann Oncol. 2011 Aug;22(8):1828-33. doi: 10.1093/annonc/mdq696. Epub 2011 Feb 2. PMID 21289369
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6181036&StudyName=A%20Treatment%20Protocol%20for%20Patients%20with%20Gastrointestinal%20Stromal%20Tumor%20%28GIST%29%20who%20May%20Derive%20Benefit%20from%20Treatment%20with%20SU011248%20%20